CLINICAL TRIAL: NCT04395859
Title: Collateral Damage From the COVID-19 Pandemic Observed in Patients Treated With Intravitreal Injections (IVT) of Anti-angiogenic Agents
Acronym: COVIDIV
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MMT_2020_15
Record Dates: First submitted 2020-05-18; First posted 2020-05-20 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Age Related Macular Degeneration; Diabetic Macular Edema; Retinal Vein Occlusion
Keywords: Intravitreal Injections; Anti-angiogenics; COVID19
MeSH Terms: conditions — Macular Degeneration; Retinal Vein Occlusion; COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with IVT before COVID19 pandemia: Treatment started at least 6 months before the French confinement for COVID19 (15th march 2020)
  Interventions: Procedure: Questionnaire; Other: Data collection up to 1 year

INTERVENTIONS:
Procedure: Questionnaire — At inclusion : Questionnaire collecting data concerning the interruption of IVT treatment
Other: Data collection up to 1 year — Data collection up to 1 year after resumption of follow-up: visual acuity, OCT : optical coherence tomography, IVT treatment, complications

SUMMARY:
In patients treated for exudative age-related macular degeneration (AMD), diabetes, retinal venous occlusion (OVR), or other conditions causing macular edema, treatments with anti-angiogenic intravitreal injections (IVT) are widely used both for their anti-angiogenic action. Patients often have injections for many years, sometimes monthly or every 2 months.

The discontinuation of treatment with repeated injections of anti-angiogenic agents, linked to the COVID-19 coronavirus pandemic will potentially impact the visual acuity, the ophthalmological state and the quality of life of the patients concerned, therefore it is relevant to analyze the consequences the breakdown of usual care in this population.

ELIGIBILITY:
Inclusion Criteria:

* Ocular pathology requiring repeated IVT treatment of anti-angiogenic drugs (exudative AMD, diabetic macular edema or secondary to retinal venous occlusion ...)
* Beginning of IVT treatment repeated before 10/01/2019 (6 months before the start of French confinement)

Exclusion Criteria:

* Refusal to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated with repeated IVT treatment of anti-angiogenic drugs
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Change of visual acuity in patients treated with repeated IVT anti-angiogens during the COVID-19 epidemic | Baseline (Before confinement) and 6 months after resumption of follow-up
  Change from baseline (last visual acuity before confinement) and visual acuity 6 months after resumption of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Martine MAUGET FAYSSE, MD, Principal Investigator — Fondation Adolphe de Rothschild
Locations (4):
- France (4):
  - Centre Pôle Vision du val d'Ouest, Écully
  - Fondation Adolphe de Rothschild, Paris
  - Hôpital Lariboisière, Paris
  - Centre ophtalmologique Maison Rouge, Strasbourg

REFERENCES:
- [Derived] Sukkarieh G, Bonnin S, Azar G, Lafolie J, Alonso AS, Erol O, Pineau J, Villain H, Guillaume J, Auge E, Mingou A, Lejoyeux R, Vasseur V, Mauget-Faysse M. Outcome of Patients Treated by Intravitreal Injections During the COVID-19 Lockdown: An Institutional Experience. Curr Eye Res. 2023 Jul;48(7):683-689. doi: 10.1080/02713683.2023.2200564. Epub 2023 Apr 12. PMID 37024478